CLINICAL TRIAL: NCT00382213
Title: A Randomized, Double Blind Study To Compare The Effects Of Olmesartan Medoxomil Versus Placebo In Patients With Established Atherosclerosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 866-422 AIMS
Record Dates: First submitted 2006-09-27; First posted 2006-09-28 (Estimated); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Atherosclerosis
MeSH Terms: conditions — Atherosclerosis | interventions — Olmesartan Medoxomil

INTERVENTIONS:
Drug: Olmesartan medoxomil
Drug: Placebo

SUMMARY:
The purpose of this study is to determine the efficacy of treatment with olmesartan medoxomil, an Angiotensin Receptor Blocker, compared to placebo on the blood levels of surrogate markers of vascular inflammation for atherosclerotic disease. Patients will be randomized to receive either olmesartan medoxomil or placebo for one year.

ELIGIBILITY:
Inclusion Criteria:

* Males or Females age less than or equal to 18
* TEE-defined Grade III or IV atherosclerotic disease of the thoracic aorta documented within the previous 90 days, or established atherosclerotic disease of the lower extremities as demonstrated by:

  * a history of lower extremity peripheral vascular surgery for obstructive atherosclerotic disease, or
  * a history of lower extremity peripheral arterial angioplasty for obstructive atherosclerotic disease, or
  * a history of lower extremity amputation secondary to atherosclerotic disease, or
  * an ABI <0.90 within the previous 90 days, or
  * a history of claudication in patients with documented coronary artery disease (i.e., history of myocardial infarction, coronary revascularization, or coronary angiography demonstrating at least one obstructive coronary lesion with a 50% or greater stenosis).

Exclusion Criteria:

* Women of childbearing age who do not agree to utilize protocol approved contraceptive methods.
* Average pre-dose SBP < 100 or DBP < 60.
* Patients with any serious disorder including cardiovascular (ventricular arrhythmias, valvular disease or implantable defibrillator), renal, pulmonary, hepatic, gastrointestinal, endocrine/metabolic (excluding patients with controlled diabetes mellitus), hematologic/oncologic (including an active malignancy other than basal cell carcinoma or non-metastatic prostate cancer), neurologic, and psychiatric diseases.
* Patients with a history of MI, PTCA, CABG, heart failure, CVA or TIA within the last 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210
Dates: Start 2000-06; Study Completion 2004-12

PRIMARY OUTCOMES:
The primary endpoint for the determination of efficacy will be a composite of
ten circulating surrogate markers of atherosclerosis for vascular inflammation.
The surrogate markers of vascular inflammation to be used will include
C-reactive protein, MCP-1, M-CSF, VCAM-1, TNFα, IL-1, E-Selectin, ICAM-1, IL-6
and MMP-9.

SECONDARY OUTCOMES:
Individual circulating surrogate markers of atherosclerosis listed above
(C-reactive protein, MCP-1, M-CSF, VCAM-1, TNFα, IL-1, E-Selectin, ICAM-1,
IL-6 and MMP).
Serum levels of TGF-β, PDGF, HGF, and PAI-1.
The ratio of reduced to oxidized glutathione in the plasma as an indicator
of oxidative stress (GSH/GSSG ratio).
Composite of adhesion markers (VCAM-1, E-selectin, and ICAM-1).
Composite of chemoattractant markers (MCP-1, M-CSF).
Composite of Growth Factor Markers (PDGF, HGF, TGF-β).
Assessment of atherosclerotic disease severity of the thoracic aorta as
determined by transesophageal echocardiography (TEE) in patients enrolled
on the basis of TEE-defined aortic atherosclerosis.
Assessment of atherosclerotic disease severity of the peripheral arteries
of the lower extremities as determined by the ankle brachial index (ABI).
Endothelial function as determined by brachial artery diameter responses to
hyperemic flow.